CLINICAL TRIAL: NCT07295847
Title: A Phase 1b, Open-label, Multi-cohort Study of AZD0120, an Autologous CD19/BCMA Targeting Chimeric Antigen Receptor T-cell, in Adults With Autoimmune Diseases
Brief Title: A Study of AZD0120 in Autoimmune Diseases
Acronym: AURORA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8318C00001; 29707 (Other: IND)
Record Dates: First submitted 2025-10-16; First posted 2025-12-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Rheumatoid Arthritis
Keywords: Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Rheumatoid Arthritis; CAR-T; BCMA; CD19
MeSH Terms: conditions — Scleroderma, Systemic; Myositis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Multi-indication cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD0120 Regimen 1 (Experimental): Participants will receive an infusion of AZD0120 Regimen 1.
  Interventions: Biological: AZD0120
- AZD0120 Regimen 2 (Experimental): Participants will receive an infusion of AZD0120 Regimen 2.
  Interventions: Biological: AZD0120

INTERVENTIONS:
Biological: AZD0120 — CD19/BCMA Autologous CAR T-cell therapy product
  Other Names: GC012F

SUMMARY:
This trial is a Phase 1b, open-label, multi-center, clinical study of AZD0120, a BCMA/CD19 dual targeting CAR+ T-cell therapy, to evaluate the safety and tolerability in adult participants with systemic sclerosis (SSc), idiopathic inflammatory myopathies (IIM), or difficult-to-treat rheumatoid arthritis (D2T RA).

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multi-center, multi-cohort clinical study of AZD0120, a CD19/BCMA dual CAR T-cell therapy, to evaluate the safety in adult participants with systemic sclerosis (SSc), idiopathic inflammatory myopathies (IIM), or difficult-to-treat rheumatoid arthritis (D2T RA) for determination of the recommended phase 2 dose for each disease cohort. Approximately 9-12 participants will be evaluated per disease cohort.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Adequate physiological function and reserve at screening.
* Able to comply with recommended medication washout period.
* Participants who are suitable for the study as determined by medical evaluation and at the discretion of the investigator.
* Willingness to remain on/start appropriate, highly effective methods of birth control or other acceptable criteria.

Exclusion Criteria:

* BMI at screening < 18 or > 35kg/m2.
* Any prior CAR T exposure.
* Unable or unwilling to remain within proximity (~2 hours travel time) of the administering investigational site for the first 28 days post study drug administration.
* Received a bone marrow or solid organ transplant at any time or on an active transplant waiting list.
* Received any investigational drug within ≥ 5 half-lives or 4 weeks, whichever is longer, prior to screening.
* Has certain heart conditions that could make it unsafe or unsuitable to take part in the study.
* Requirement for supplemental oxygen at rest (except at night for sleep apnea) or mechanical ventilation.
* Uncontrolled hypertension (> 160/100 mmHg) or symptomatic hypertension.
* Any central nervous system disease that may impact participants safety in the investigator's opinion.
* Other concurrent autoimmune or autoinflammatory disease. Certain autoimmune/autoinflammatory diseases may be included after discussion with the medical monitor.
* Evidence of clinically significant bleeding or active bleeding conditions within 90 days before screening
* History of malignancy or ongoing treatment for prior malignancy. Certain malignancies may be excepted.
* Known genetic inborn error of immunity and/or primary immunodeficiency.
* Active viral, bacterial, or fungal infection, or any ongoing infection that requires systemic antimicrobial therapy in the 4 weeks prior to screening.
* Seropositive for HIV.
* Active viral hepatitis are excluded.
* Active syphilis, positive for Treponema pallidum antibody.
* Vaccinated with live, attenuated vaccine within 4 weeks prior to apheresis or lymphodepletion.
* Not up-to-date on vaccinations per local/national health authority or institutional guidelines for immune-compromised individuals.
* Known life threatening allergies, hypersensitivity, or intolerance to AZD0120 or its excipients, including dimethyl sulfoxide.
* Contraindications or hypersensitivity to fludarabine and cyclophosphamide.
* Major surgery, or has surgery planned during the study.
* Pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 1 year after receiving study treatment (whichever is later).
* Plans to father a child while enrolled in this study or within 1 year after receiving study treatment (whichever is later).
* Any issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to provide informed consent or any condition in the opinion of the investigator, participation would not be in the best interest of the participant.

Other protocol-defined eligibility criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2028-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants and severity of dose limiting toxicities (DLTs) and treatment-emergent adverse events (TEAEs) | 1 year
  Incidence and severity of DLTs and TEAEs to evaluate the safety of AZD0120 and to confirm the recommended Phase 2 dose (RP2D) in each indication SSc, IIM, or RA

SECONDARY OUTCOMES:
Cellular Kinetics - Cmax | 1 year
  The maximum concentration of CAR T cells achieved in the body.
Cellular Kinetics - Tmax | 1 year
  The time point at which the Cmax is reached
Cellular Kinetics - AUC | 1 year
  The area under the concentration-time curve, which represents the total drug exposure over a specific period.
Cellular Kinetics - t½λz | 1 year
  The terminal elimination half-life.
Cellular Kinetics - Clast | 1 year
  The last observed quantifiable concentration of CAR T-cells.
Cellular Kinetics - Tlast | 1 year
  The time to last quantifiable concentration.
Cellular Kinetics - AUClast | 1 year
  The area under the concentration-time curve to the last measurable concentration.
Anti-drug antibodies (ADA) developed against AZD0120 from baseline | 1 year
  Humoral immunogenicity assessment of AZD0120 in participants with SSc, IIM, or RA.
Proportion of participants with detectable replication competent lentivirus (RCL) at pre-specified post infusion timepoints. | 1 year
  Incidence of vector-derived RCL in participant receiving AZD0120.
Change from baseline in the Disease Activity Score (DAS) 28-C-reactive protein (CRP). The DAS28-CRP is a measure from 0-10 with higher scores indicating greater disease activity. | 1 year
  Disease activity measures in RA participants.
Change from baseline in modified Rodnan Skin Score (mRSS). The mRSS is a measure of skin thickness with a range of 0-51 with higher scores indicating more severe disease. | 1 year
  Disease activity measures in SSc participants.
Change from baseline in the total improvement score (TIS). The TIS ranges from 0-100 with higher scores indicating greater improvement. | 1 year
  Disease activity measures in IIM participants.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - Research Site, Tucson, Arizona
  - Research Site, Stanford, California
  - Research Site, Chicago, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Darlinghurst
  - Research Site, Waratah
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Mainz Am Rhein
  - Research Site, Würzburg
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, Edinburgh
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/